CLINICAL TRIAL: NCT02311777
Title: Effects of Pre-operative Pregabalin and Ketamine to Prevent Development of Phantom Pain in Patients Undergoing Lower Extremity Amputation
Brief Title: Pre-operative Pregabalin and Ketamine to Prevent Phantom Pain
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Preoperative period is very short time
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dawood Nasir, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: STU 092014-050
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Phantom Pain
MeSH Terms: conditions — Phantom Limb | interventions — Pregabalin; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin-ketamine (Active Comparator): Pregabalin and ketamine will be given preoperative period
  Interventions: Drug: Pregabalin; Drug: Ketamine
- Placebo (Placebo Comparator): Placebo will be given preoperative period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin will be given orally during preoperative period
  Other Names: Lyrica
  Arms: Pregabalin-ketamine
Drug: Ketamine — Ketamine will be given on the surgery day before the anesthesia induction
  Other Names: Ketamine hydrocloride
  Arms: Pregabalin-ketamine
Drug: Placebo — Placebo will be given orally during preoperative period
  Other Names: Placebo pregabalin/placebo ketamine
  Arms: Placebo

SUMMARY:
Phantom limb pain (PLP) is as painful sensations located to the missing limb and classified as neuropathic pain. In the United States, an estimated 1.7 million patients have undergone limb amputation, and 60% to 80% of these patients develop PLP (1-2) and it is usually resistant to a wide variety of treatments (1-4). Three factors may contribute to the development of persistent, post-amputation PLP by inducing central sensitization at different times relative to surgery: pre-amputation pain, noxious intraoperative stimuli, and acute postoperative pain (5-7).

Investigators hypothesis that pre-amputation period could be important in eliminating Phantom Limb Pain (PLP) in the patients in whom cortical reorganization is not yet established. The reduction of pre-operative pain and prevention of formation of pain memories may eliminate development of PLP by using dual networks treatment strategy. This Phase III, randomized, double-blind, placebo-controlled study is designed to evaluate the efficacy of pre-operative pregabalin (lyrica) and ketamine in eliminating phantom limb pain in patients undergoing lower limb amputation.

DETAILED DESCRIPTION:
Patients undergoing unilateral lower extremity amputation (n=30) will be randomized in this double blind parallel placebo control clinical trial to evaluate the efficacy of pre-operative pregabalin (lyrica) and ketamine in eliminating phantom limb pain. Patient will receive either pregabalin and ketamine treatment (Group 1) or placebo (Group 2) during pre-operative period approximately 4 days (2-4 days).

Patients will be identified during their anesthesia preoperative clinic or orthopedic inpatient unit (Parkland Hospital or UT Southwestern University Hospital) for the eligibility. Data base (EPIC) will also be used for prescreening of potential subject by reviewing clinic visit daily schedule or operating room schedule. Then patients chart will be reviewed for initial data collection to determine the eligibility of potential subjects with the use of a HIPAA waiver form. Eligible subject will be approached by the study PI, investigators, or research coordinator and written consent obtained prior to any study procedures.

A pregnancy test will be performed before the preoperative treatment start for women in child-bearing age: exceptions include surgically sterile women or women with medically confirmed menopause. Women with a positive pregnancy test or who report unprotected heterosexual sex since their previous menses or not currently using and/or willing to use a medically approved form of contraception (e.g., birth control pill) will not enrolled to the study.

Pain will be documented using the visual analog pain score (0=no pain, 10=worst imaginary pain) during preoperative period before the treatment and daily on pain diary and on the day of surgery and during postoperative period at PACU, 24 and 48 hrs. and long-term follow-up 1, 3, and 6 months after the surgery.

Total opioid dose over the 48-h study period will be documented as PCA pump morphine consumption for postoperative first 24 hrs. and postoperative oral opioid usage for 48 hrs. after surgery. Patients will receive a standard general anesthetic for their surgery and postoperative standard of care pain treatment similar to all patients. Study does not limit standard post-operative pain medication.

Long-term analgesic success will be evaluated at 1, 3, and 6 months after surgery. At follow-up period, a pain diary will be used for the patients' self-assessment on pain occurrence, intensity, duration for phantom and stump pain, and documentation of oral analgesic usage. Analgesic medication use and daily pain scores will be documented on pain diary for 1 month period following surgery. At first follow-up visit, patient will be seen in Pain Clinic 1 month after the surgery. Patient will be called from home 3 and 6 months after the surgery for long-term follow-up.

At all-time points, the Self-Rating Depression Scale will be used to assess depression and the patients will complete the Pain-Related Self-Statement Scale (PRSS).

The duration of the involvement in the study will be 6 months.

Randomization:

This is randomized double-blinded placebo controlled clinical trial. Investigational Drug Pharmacy (IDS) will randomize subjects either treatment group or placebo. IDS will dispense the drugs/placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Ager 18-65 years old
2. Unilateral lower-limb amputations
3. Able to understand study procedures
4. If on opioids, patient should be on a stable dose for at least one week prior to enrolment.
5. Subject with normal renal function (CrCI > 60 mL/min).

Exclusion Criteria:

1. Cases with only digits amputation
2. Current or recent history of alcohol and drug abuse
3. Concomitant use of CYP 3A4 medications
4. Unstable hypertension
5. Abnormal EKG
6. Increased intracranial pressure currently or in the past six months
7. Increased intraocular pressure currently or in the past six months
8. Liver disease or AST/ALT ≥ 3 ULN or total bilirubin >2 x ULN
9. Poorly controlled psychiatric illness.
10. A history of seizure
11. Using other anticonvulsant drug
12. Renal impairment as determined by clinically significant labs
13. Women of childbearing age who either has:

    1. A positive pregnancy test
    2. Unprotected heterosexual sex since their previous menses or;
    3. Not currently using and/or willing to use a medically approved form of contraception (e.g., birth control pill)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-09-20 (Estimated); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Pain Scores (VAS) | Postoperaive 6 months
  Pain will be evaluated immediate postoperative period and 6 months after surgery

SECONDARY OUTCOMES:
Oral analgesic consumption | 1 months after surgery
  Amounts of rescue analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Dawood H Nasir, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health Hospital System, Dallas, Texas
  - UTSW, Parkland Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No